CLINICAL TRIAL: NCT01949168
Title: Phase 2a Study of Boceprevir for the Treatment of Genotype 6 Hepatitis C
Brief Title: A Pilot Study of Boceprevir for the Treatment of Genotype 6 HCV
Acronym: HCV-6
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St Vincent's Hospital Melbourne (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Alexander Thompson, Head of Hepatology Research, St Vincent's Hospital Melbourne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCV-6 study
Record Dates: First submitted 2013-09-04; First posted 2013-09-24 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Boceprevir triple therapy with 5-day lead in (Active Comparator): Victrelis® (boceprevir) 800mg by mouth, TID (200 mg tablets) for 5 days, followed by boceprevir plus • Peg-Intron® (peginterferon-α-2b), 1.5ug/kg sc injection plus • Rebetol® (ribavirin), 1000/1200mg, by mouth daily for 24 weeks. In patients who achieve an undetectable plasma HCV RNA level at week 4 of triple therapy (week 5 from baseline), and maintain an undetectable plasma HCV RNA at week 20 of triple therapy (week 21 from baseline), treatment will stop at week 25. Patients who have a detectable plasma HCV RNA at week 4 of triple therapy, but an undetectable plasma HCV RNA at week 20, will continue a with follow-on peginterferon-α-2b plus ribavirin for a further 23 weeks (stopping at week 48).
  Interventions: Drug: Victrelis® (boceprevir) 800mg by mouth, TID (200 mg tablets); Drug: Peg-Intron® (peginterferon-α-2b), 1.5ug/kg sc injection; Drug: Rebetol® (ribavirin), 1000/1200mg by mouth daily
- Boceprevir triple therapy (Active Comparator): Victrelis® (boceprevir) 800mg by mouth, TID (200 mg tablets) plus Peg-Intron® (peginterferon-α-2b), 1.5ug/kg sc injection and Rebetol® (ribavirin), 1000/1200mg, by mouth daily for 24 weeks. In patients who achieve an undetectable plasma HCV RNA level at week 4 of triple therapy, and maintain an undetectable plasma HCV RNA at week 20 of triple therapy, treatment will stop at week 24. Patients who have a detectable plasma HCV RNA at week 4 of triple therapy, but an undetectable plasma HCV RNA at week 20, will continue a with follow-on peginterferon-α-2b plus ribavirin for a further 24 weeks (stopping at week 48).
  Interventions: Drug: Victrelis® (boceprevir) 800mg by mouth, TID (200 mg tablets); Drug: Peg-Intron® (peginterferon-α-2b), 1.5ug/kg sc injection; Drug: Rebetol® (ribavirin), 1000/1200mg by mouth daily
- Standard of Care (Active Comparator): 48 weeks of Peg-Intron® (peginterferon-α-2b), 1.5ug/kg sc injection and Rebetol® (ribavirin), 1000/1200mg by mouth daily (200mg tablets)
  Interventions: Drug: Peg-Intron® (peginterferon-α-2b), 1.5ug/kg sc injection; Drug: Rebetol® (ribavirin), 1000/1200mg by mouth daily

INTERVENTIONS:
Drug: Victrelis® (boceprevir) 800mg by mouth, TID (200 mg tablets)
  Arms: Boceprevir triple therapy; Boceprevir triple therapy with 5-day lead in
Drug: Peg-Intron® (peginterferon-α-2b), 1.5ug/kg sc injection
Drug: Rebetol® (ribavirin), 1000/1200mg by mouth daily

SUMMARY:
The purpose of this study is to evaluate the antiviral efficacy of Boceprevir-based therapy for the treatment of genotype 6 chronic hepatitis C infection.

Boceprevir has recently been approved for the treatment of genotype 1 chronic hepatitis C infection. Recent in vitro studies suggest similar efficacy against genotype 6 chronic hepatitis C infection.

The investigators therefore hypothesise that:

i) Boceprevir is a potent inhibitor of genotype 6 hepatitis C replication in vivo.

ii) Boceprevir in combination with pegylated interferon-alpha and ribavirin for 24 weeks will cure a high proportion of patients chronically infected with genotype 6 chronic hepatitis C infection.

DETAILED DESCRIPTION:
Genotype 6 HCV (HCV-6) is common in parts of South-East Asia, in particular Vietnam. There is a small but growing population of immigrant patients with chronic HCV-6 in Australia. The current standard-of-care treatment (SOC) for chronic HCV-6 infection is peg-interferon-α (PEG-IFN) and ribavirin (RBV) therapy for 48 weeks. The available data evaluating treatment outcome suggests that SVR rates are intermediate between those of HCV-1 and HCV-2/3. There is a medical need for novel therapies that might increase SVR rates and/or allow shortened treatment duration.

Boceprevir is a novel HCV NS3 protease inhibitor, and boceprevir-based triple therapy has recently been approved for the treatment of HCV-1. Boceprevir also appears to have some antiviral effect against HCV-2 and HCV-3 in vivo. Boceprevir has not been used to treat patients with chronic HCV-6 infection. Recent in vitro data have demonstrated that boceprevir has an antiviral effect against HCV-6.

The investigators are therefore undertaking an investigator-initiated proof-of-concept pilot study of boceprevir-based therapy for the treatment of patients chronically infected with HCV-6.

The study population will consist of a representative group of 30 adult patients who are chronically infected with genotype 6 HCV. All patients will be of Asian background, will be non-cirrhotic, and will carry a "good response" IL28B genotype (C/C for rs12979860). The patients will be recruited from the outpatient clinics of 4 Hepatology units in Melbourne, Australia, represented by the principal and associate investigators.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age
* Asian background
* HCV treatment-naïve.
* Chronic HCV infection is defined as one of the following:
* Positive for anti-HCV antibody (Ab) or HCV RNA at least 6 months before Screening, and positive for HCV RNA and anti-HCVAb at the time of Screening; or
* Positive for anti-HCV Ab and HCV RNA at the time of Screening with a liver biopsy consistent with chronic HCV infection (or a liver biopsy performed prior to enrollment with evidence of chronic hepatitis C disease).
* Screening laboratory result indicating HCV genotype 6-infection (HCV-6).
* Plasma HCV RNA level > 10,000 IU/mL at Screening.
* IL28B C/C genotype (rs12979860)
* Per local standard practice, documented results of one of the following:
* A liver biopsy within 24 months prior to or during screening demonstrating the absence of cirrhosis, e.g., a METAVIR Score of 3 or less, Ishak score of 4 or less; or
* A screening FibroTest score of ≤ 0.72 and Aspartate Aminotransferase to Platelet Ratio Index (APRI) ≤ 2; or
* A screening FibroScan result of < 9.6 kPa.
* Subjects with a non-qualifying Fibrotest/APRI or Fibroscan result may only be enrolled if they have a qualifying liver biopsy preformed within 24 months prior to or during screening.
* Candidate for PEG/RBV therapy
* Body mass index (BMI) between 18 and 36 kg/m2
* Agree to use two highly effective methods of avoiding contraception for the duration of the study and for 7 months after the last dose study medication. Females of childbearing potential must have negative pregnancy test at Screening and Baseline
* Provide written informed consent to participate in the study.
* Subjects must have the following laboratory parameters at Screening:
* ALT ≤ 10 × the upper limit of normal (ULN)
* AST ≤ 10 × ULN
* Hemoglobin ≥ 12 g/dL
* White blood cell count ≥ 2,500 cells/μL
* Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
* Platelets ≥ 90,000/mm3
* Prothrombin time ≤ 1.5 × ULN
* Albumin > 3 g/dL
* Direct (conjugated) bilirubin < ULN
* Thyroid stimulating hormone (TSH) ≤ ULN
* Creatinine clearance (CLcr) ≥ 50 mL/min, as calculated by the Cockcroft-Gault equation

Exclusion Criteria:

* Non-genotype 6 HCV infection, or evidence of mixed genotype HCV infection
* IL28B C/T or T/T polymorphism (rs12979860)
* Any current or past clinical evidence of cirrhosis such as ascites or esophageal varices, or prior biopsy showing cirrhosis, e.g., a Metavir Score of >3 or Ishak score of > 4.
* Exceed defined thresholds for key laboratory parameters at Screening.
* Females who are pregnant or plan to become pregnant, or breastfeeding, or males whose partners are pregnant or planning to become pregnant within 7 months (or per local RBV label) after their last dose of study drug.
* Positive test result for Hepatitis B surface antigen (HBsAg) or anti-Human immunodeficiency virus antibody (HIV Ab).
* Diagnosis of autoimmune disease, decompensated liver, disease, poorly controlled diabetes mellitus, significant psychiatric illness, severe chronic obstructive pulmonary disease (COPD), hepatocellular carcinoma or other malignancy (with exception of certain skin cancers), hemoglobinopathy, retinal disease, or are immunosuppressed
* Subjects with current use of amphetamines, cocaine, opiates (e.g., morphine, heroin), or ongoing alcohol abuse are excluded. Subjects on stable methadone maintenance treatment for at least 6 months prior to Screening may be included into the study.
* Use of prohibited concomitant medications two weeks prior to baseline through the end of treatment, as defined by the product label.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Early viral kinetics | Day 5
  Determined by plasma HCV RNA quantification at frequent time points - baseline, day 1, 2, 3, 4 and 5

SECONDARY OUTCOMES:
Rates of virological response | Day 3, 5, week 2, week 4, week 12 and end of treatment (week 24 or week 48)
  Percentage of patients with undetectable plasma HCV RNA) at different time-points
Number of patients eligible for Response Guided Therapy | Week 4 and week 20
  Patients in Arm A and B randomised to received boceprevir-based triple therapy who achieve an undetectable HCV PCR at week 4 and week 20 are eligible for 24 weeks of therapy, vs. 48 weeks of therapy
Rates of virological breakthrough | Week 4, week 20, week 24, week 48, week 60
  Defined by an increase in HCV RNA > 1 log10 IU/mL from nadir, or HCV RNA increase to > 100 IU/mL in patients who had previously reached an undetectable HCV RNA, and confirmed by 2 consecutive samples < 4 weeks apart.
Rates of SVR12 and relapse | Week 48 and Week 60
  SVR 12 - Number of patients who achieve an undetectable HCV PCR 12-weeks post treatment Relapse - Number of patients who have an undetectable HCV PCR at the end of treatment but detectable HCV PCR 12-weeks post treatment
Rates of anaemia on treatment | Day 0, 1, 2, 3, 4, 5, then monthly up to week 48 of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Thompson, MBBS, Principal Investigator — St Vincent's Hospital Melbourne
Locations (4):
- Australia (4):
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - St Vincent's Hospital, Fitzroy, Victoria
  - Western Hospital, Footscray, Victoria

REFERENCES:
- [Background] Sievert W, Altraif I, Razavi HA, Abdo A, Ahmed EA, Alomair A, Amarapurkar D, Chen CH, Dou X, El Khayat H, Elshazly M, Esmat G, Guan R, Han KH, Koike K, Largen A, McCaughan G, Mogawer S, Monis A, Nawaz A, Piratvisuth T, Sanai FM, Sharara AI, Sibbel S, Sood A, Suh DJ, Wallace C, Young K, Negro F. A systematic review of hepatitis C virus epidemiology in Asia, Australia and Egypt. Liver Int. 2011 Jul;31 Suppl 2:61-80. doi: 10.1111/j.1478-3231.2011.02540.x. PMID 21651703
- [Background] Dev AT, McCaw R, Sundararajan V, Bowden S, Sievert W. Southeast Asian patients with chronic hepatitis C: the impact of novel genotypes and race on treatment outcome. Hepatology. 2002 Nov;36(5):1259-65. doi: 10.1053/jhep.2002.36781. PMID 12395338
- [Background] Ghany MG, Strader DB, Thomas DL, Seeff LB; American Association for the Study of Liver Diseases. Diagnosis, management, and treatment of hepatitis C: an update. Hepatology. 2009 Apr;49(4):1335-74. doi: 10.1002/hep.22759. No abstract available. PMID 19330875
- [Background] Poordad F, McCone J Jr, Bacon BR, Bruno S, Manns MP, Sulkowski MS, Jacobson IM, Reddy KR, Goodman ZD, Boparai N, DiNubile MJ, Sniukiene V, Brass CA, Albrecht JK, Bronowicki JP; SPRINT-2 Investigators. Boceprevir for untreated chronic HCV genotype 1 infection. N Engl J Med. 2011 Mar 31;364(13):1195-206. doi: 10.1056/NEJMoa1010494. PMID 21449783
- [Background] Bathgate A. Boceprevir for previously treated chronic hepatitis C virus genotype 1 infection. J R Coll Physicians Edinb. 2011 Jun;41(2):122-3. doi: 10.4997/JRCPE.2011.222. No abstract available. PMID 21677916
- [Background] Silva MO, Treitel M, Graham DJ, Curry S, Frontera MJ, McMonagle P, Gupta S, Hughes E, Chase R, Lahser F, Barnard RJ, Howe AY, Howe JA. Antiviral activity of boceprevir monotherapy in treatment-naive subjects with chronic hepatitis C genotype 2/3. J Hepatol. 2013 Jul;59(1):31-7. doi: 10.1016/j.jhep.2013.02.018. Epub 2013 Feb 27. PMID 23454058
- [Background] Ge D, Fellay J, Thompson AJ, Simon JS, Shianna KV, Urban TJ, Heinzen EL, Qiu P, Bertelsen AH, Muir AJ, Sulkowski M, McHutchison JG, Goldstein DB. Genetic variation in IL28B predicts hepatitis C treatment-induced viral clearance. Nature. 2009 Sep 17;461(7262):399-401. doi: 10.1038/nature08309. Epub 2009 Aug 16. PMID 19684573